CLINICAL TRIAL: NCT03557385
Title: Adenosine Contrast CorrELations in Evaluating RevAscularizaTION
Acronym: ACCELERATION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Acist Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00093001
Record Dates: First submitted 2018-05-18; First posted 2018-06-15 (Actual); Results first posted 2024-04-02 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Percutaneous Coronary Intervention
Keywords: Fractional Flow Reserve
MeSH Terms: interventions — Iopamidol; Adenosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- aFFR vs cFFR (Other): All subjects will receive Fractional Flow Reserve Measurements with both adenosine (aFFR) and contrast (Iopamidol) (cFFR) using the Navvus® Catheter and CVi® Contrast Delivery System
  Interventions: Drug: Iopamidol; Drug: adenosine; Device: Navvus® Catheter; Device: CVi® Contrast Delivery System

INTERVENTIONS:
Drug: Iopamidol — aFFR measurement with drug: Iopamidol (ISOVUE®-370). Subjects will receive an injector-based intracoronary bolus of contrast
  * Rate of 4 mL/sec, volume of 10 cc (left coronary system)
  * Rate of 3 mL/sec, volume of 6 cc (right coronary system).
  Other Names: Contrast Fractional Flow Reserve Measurement
Drug: adenosine — FFR measurement with drug: adenosine. Intravenous adenosine will be administered at a rate of 140 μg/kg of body weight per minute x 2 minutes
  Other Names: Adenosine Fractional Flow Reserve Measurement
Device: Navvus® Catheter — the NAVVUS RXi microcatheter will be used with a workhorse wire of the operator's choosing
Device: CVi® Contrast Delivery System — The CVi® Contrast Delivery System will be used to deliver the contrast medium

SUMMARY:
The purpose of this study is to compare FFR measurements done with adenosine to FFR measurements done with contrast, where the contrast is injected using the ACIST CVi automated contrast injector.

The ACCELERATION study will support a safer approach to FFR for patients by potentially reducing toxic drug exposure (adenosine). The 2 main objectives of the study are:

1. Perform a methods comparison between cFFR and the reference standard aFFR, where cFFR is performed using an automated injector with a standardized volume and rate of delivery of contrast with known osmolality.
2. Evaluate the association between final post-PCI FFR and long-term clinical outcomes. The long-term clinical outcomes will include TVR and composite MACE (death, MI, and TVR) at 30 days and 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Have the capacity to understand and sign an informed consent or have a legally authorized representative (LAR) that can understand and sign an informed consent prior to initial arteriotomy access
2. Age > 18 years of age at the time of signing the informed consent
3. Clinically stable and undergoing non-emergent cardiac catheterization for appropriate indications
4. Willing to be contacted by telephone at 30 days (if no standard of care visit) and at 1 year with chart review for events.
5. Target vessel with an intermediate lesion of 40-70% stenosis by angiographic assessment (a visual estimation by the operator). Serial lesions, diffuse disease, or ostial lesions ("all-comer" lesions) are acceptable if the operator would normally perform FFR and proceed with PCI (or other revascularization) if positive.

Exclusion Criteria:

1. Any condition associated with a life expectancy of less than 1 year
2. Participation in another clinical study using an investigational agent or device within the past 3 months
3. Ejection fraction ≤ 35%
4. Creatinine ≥ 2
5. Severe valvular heart disease
6. Decompensated acute diastolic or systolic heart failure
7. Bronchospastic chronic obstructive pulmonary disease or other intolerance to adenosine
8. ST-segment elevation myocardial infarction culprit lesion or lesions with any thrombus burden after diagnostic angiography
9. Lesions with severe calcification after diagnostic angiography
10. Lesions in a target vessel supplied by a patent graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Swaminathan, MD, Principal Investigator — DCRI
Locations (5):
- United States (5):
  - Long Beach VA, Long Beach, California
  - Mercy Hospital, Coon Rapids, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Durham VA, Durham, North Carolina
  - Vanderbilt, Nashville, Tennessee

REFERENCES:
- [Derived] Swaminathan RV, Marquis-Gravel G, Boivin-Proulx LA, Benjamin DK, Rikhi A, Raveendran G, Chambers JW, Seto AH, Bagai J, White R, Gutierrez JA, Povsic TJ, Rao SV, Krucoff MW. Adenosine Contrast Correlations in Evaluating Revascularization: The (ACCELERATION) Study. Circ Cardiovasc Interv. 2025 Jun;18(6):e015240. doi: 10.1161/CIRCINTERVENTIONS.125.015240. Epub 2025 Apr 24. PMID 40270240

RESULTS

PARTICIPANT FLOW:
Groups:
- aFFR and cFFR: All subjects will receive Fractional Flow Reserve Measurements with both adenosine (aFFR) and contrast (Iopamidol) (cFFR) using the Navvus® Catheter and CVi® Contrast Delivery System
  Iopamidol: aFFR measurement with drug: Iopamidol (ISOVUE®-370). Subjects will receive an injector-based intracoronary bolus of contrast
  * Rate of 4 mL/sec, volume of 10 cc (left coronary system)
  * Rate of 3 mL/sec, volume of 6 cc (right coronary system).
  adenosine: FFR measurement with drug: adenosine. Intravenous adenosine will be administered at a rate of 140 μg/kg of body weight per minute x 2 minutes
  Navvus® Catheter: the NAVVUS RXi microcatheter will be used with a workhorse wire of the operator's choosing
  CVi® Contrast Delivery System: The CVi® Contrast Delivery System will be used to deliver the contrast medium
Period: aFFR
Arm/Group | aFFR and cFFR
Started | 201
Completed | 201
Not Completed | 0
Period: cFFR
Arm/Group | aFFR and cFFR
Started | 201
Completed | 201
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analyses include all participants who completed aFFR and cFFR measurements.
Groups:
- aFFR vs cFFR: All subjects will receive Fractional Flow Reserve Measurements with both adenosine (aFFR) and contrast (Iopamidol) (cFFR) using the Navvus® Catheter and CVi® Contrast Delivery System
  Iopamidol: aFFR measurement with drug: Iopamidol (ISOVUE®-370). Subjects will receive an injector-based intracoronary bolus of contrast
  * Rate of 4 mL/sec, volume of 10 cc (left coronary system)
  * Rate of 3 mL/sec, volume of 6 cc (right coronary system).
  adenosine: FFR measurement with drug: adenosine. Intravenous adenosine will be administered at a rate of 140 μg/kg of body weight per minute x 2 minutes
  Navvus® Catheter: the NAVVUS RXi microcatheter will be used with a workhorse wire of the operator's choosing
  CVi® Contrast Delivery System: The CVi® Contrast Delivery System will be used to deliver the contrast medium
Arm/Group | aFFR vs cFFR
Number analyzed (Participants) | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.22 (8.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 171
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 195
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 182
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 201

OUTCOME MEASURES:

1. Primary Outcome: Comparison Between Contrast Fractional Flow Reserves (cFFR) and Adenosine Fractional Flow Reserves (aFFR)
Description: FFR is the ratio between the maximal myocardial flow measured in a diseased coronary artery and the theoretical maximal blood flow in the same territory in the absence of the stenosis, measured using adenosine induced hyperemia (aFFR) or contrast induced hyperemia (cFFR). Contrast FFR is being compared to the gold-standard adenosine FFR. An aFFR equal or less than 0.80 is the gold-standard cut-off to benefit from intervention. Reported as the percentage of agreement between aFFR and cFFR.
Time Frame: Baseline
Population: All subjects received Fractional Flow Reserve Measurements with both adenosine (aFFR) and contrast (Iopamidol) (cFFR) using the Navvus® Catheter and CVi® Contrast Delivery System. The FFR tracings of 217 lesions from 201 participants were assessed for quality and validity by the Fractional Flow Reserve Core Lab. After qualitative review, 192 FFR pairs were included in the analysis.
Measure: Number (95% Confidence Interval); unit: proportion of lesions with agreement
Units Other Than Participants: lesions
Groups:
- aFFR vs cFFR: All subjects will receive Fractional Flow Reserve Measurements with both adenosine (aFFR) and contrast (Iopamidol) (cFFR) using the Navvus® Catheter and CVi® Contrast Delivery System Iopamidol: aFFR measurement with drug: Iopamidol (ISOVUE®-370). Subjects will receive an injector-based intracoronary bolus of contrast Rate of 4 mL/sec, volume of 10 cc (left coronary system) Rate of 3 mL/sec, volume of 6 cc (right coronary system). adenosine: FFR measurement with drug: adenosine. Intravenous adenosine will be administered at a rate of 140 μg/kg of body weight per minute x 2 minutes Navvus® Catheter: the NAVVUS RXi microcatheter will be used with a workhorse wire of the operator's choosing CVi® Contrast Delivery System: The CVi® Contrast Delivery System will be used to deliver the contrast medium
Arm/Group | aFFR vs cFFR
Number analyzed (Participants) | 178
Number analyzed (lesions) | 192
proportion of lesions with agreement | 0.8922 [0.8403 to 0.9441]

2. Primary Outcome: Qualitative Method Comparison Between Contrast Fractional Flow Reserves and Adenosine Fractional Flow Reserves
Description: The qualitative method comparison assesses the agreement as to which lesion is flow limiting. The contrast FFR measurement that corresponds to adenosine FFR measurement value of 0.8 will be used as the cutoff value for determining whether a lesion is flow limiting for contrast FFR. Reported as the percentage of agreement between aFFR and cFFR.
Time Frame: Baseline
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of lesions with agreement
Units Other Than Participants: lesions
Arm/Group | aFFR vs cFFR
Number analyzed (Participants) | 178
Number analyzed (lesions) | 192
proportion of lesions with agreement | 0.8912 [0.8445 to 0.9379]

3. Secondary Outcome: Long-term Clinical Outcomes: Composite Major Adverse Cardiac Events (MACE: Death, MI, and TVR)
Description: (MACE: death, MI, and TVR) TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel including the target lesion.
  An MI is caused by decreased or complete cessation of blood flow to a portion of the myocardium.
Time Frame: 30 days post procedure
Population: After quality assessment, 178 patients were included in the analysis
Measure: Number; unit: Events (composite of death, MI, or TVR)
Groups:
- Per Protocol Study Population: All subjects will receive Fractional Flow Reserve Measurements with both adenosine (aFFR) and contrast (Iopamidol) (cFFR) using the Navvus® Catheter and CVi® Contrast Delivery System
Arm/Group | Per Protocol Study Population
Number analyzed (Participants) | 178
Events (composite of death, MI, or TVR) | 3

4. Secondary Outcome: Long-term Clinical Outcomes: Composite Major Adverse Cardiac Events (MACE: Death, MI, and TVR)
Description: as for outcome 3
Time Frame: 1 year post procedure
Population: After quality assessment, 178 patients were included in the analysis
Measure: Number; unit: Events (composite of death, MI, or TVR)
Arm/Group | Per Protocol Study Population
Number analyzed (Participants) | 178
Events (composite of death, MI, or TVR) | 13

ADVERSE EVENTS:
Time Frame: 1 year post procedure
Description: Adverse Event data was not collected "per arm" because aFFR and cFFR measurements were made at the same timepoints. Reported AEs include serious adverse events (SAEs) related to the NAVVUS Rxi FFR microcatheter system.
Arm/Group | aFFR vs cFFR
All-Cause Mortality (participants affected / at risk) | 7/201
Serious Adverse Events (participants affected / at risk) | 6/201
Other Adverse Events (participants affected / at risk) | 0/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | aFFR vs cFFR (N=201)
Myocardial infarction (Cardiac disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT03557385/Prot_SAP_000.pdf